CLINICAL TRIAL: NCT07047430
Title: The Airports, Air Quality, and Asthma (AAA) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Elena Austin, Assistant Professor, Environmental & Occupational Health Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00019144
Record Dates: First submitted 2025-06-04; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Asthma
Keywords: air quality; indoor air; portable air cleaner; pediatric asthma; community health workers
MeSH Terms: interventions — Air Filters

STUDY DESIGN:
Intervention Model Description: The design is a parallel group, two-arm randomized superiority trial. After enrollment, participating households are block randomized to either an intervention group or a control group in a 1:1 ratio overall and further balanced 1:1 within groups by household smoking status, defined as reported presence vs. absence of smoking household members. At the start of the trial, an indoor air cleaner is set up in the bedroom of the participating child. Air cleaners in intervention group homes are outfitted with a set of three filters (pre-filter, activated carbon filter, and HEPA filter) while those in control group homes receive an air cleaner with only a pre-filter. All households are followed for a three-month observation period that coincides with administration of the intervention.
Who Masked: Participant, Care Provider
Masking Description: Participants and CHWs are masked to intervention status. The research team, including those who attend the home visit or manage and analyze data, are not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effective portable air cleaner (HEPA) (Experimental): During the baseline home visit, a Winix 9800 air cleaner is installed in the child's bedroom and paired with data logging energy use monitor as well as air quality monitor. Households randomized to the intervention group receive an air cleaner with a pre-filter, carbon filter, and with the HEPA air filter pre-installed.
  Interventions: Device: Portable air cleaner with HEPA filter
- Control portable air cleaner (less effective). (Sham Comparator): During the baseline home visit, a Winix 9800 air cleaner is installed in the child's bedroom. In the sham group, the Winix 9800 true HEPA filter and activated carbon filter which were removed via an internal modification not visible to the user. The air cleaner still included a washable fine mesh pre-filter that captures large airborne particles. Households randomized to the sham group receive an air cleaner with only the pre-filter and without the carbon filter, and HEPA air filter.
  Interventions: Device: Less effective portable air cleaner (no HEPA)

INTERVENTIONS:
Device: Portable air cleaner with HEPA filter — The Winix 9800 is a true HEPA air cleaner that has been AHAM (Association of Home Appliance Manufacturers) Verifide® for rooms that are 500 square feet in size. The air cleaner has a washable fine mesh pre-filter that captures large airborne particles, an activated carbon filter that reduces volatile organic compounds and odors, and a true HEPA filter that captures 99.99% of airborne allergens as small as 0.003 microns in size.
  Other Names: HEPA; Portable air cleaner; Air Filter
  Arms: Effective portable air cleaner (HEPA)
Device: Less effective portable air cleaner (no HEPA) — Winix 9800 air cleaner, with data logging energy use monitor is installed in the child's bedroom. In the sham group, the Winix 9800 true HEPA filter and activated carbon filter were removed. This was an internal modification and not visible to the user. The air cleaner still included a washable fine mesh pre-filter that captures large airborne particles.
  Other Names: portable air cleaner; HEPA filter removed
  Arms: Control portable air cleaner (less effective).

SUMMARY:
For children with asthma, exposure to indoor air pollution increases the risk of a serious asthma exacerbation, which can be life-threatening. Interventions aimed at improving indoor air quality, including use of a portable air cleaner with a high-efficiency particulate air (HEPA) filter, can reduce this risk, but the effectiveness, feasibility and acceptability of HEPA air cleaners varies by setting. In collaboration with a community health worker (CHW) delivered asthma education program, the investigators are conducting a randomized clinical trial to evaluate the effectiveness of HEPA air cleaners to improve indoor air quality and child asthma health in South King County of Washington state, a vulnerable community impacted by air pollution from airports and highway traffic. Key features of the Airports, Air Quality and Asthma (AAA) design include integration of CHWs into study procedures, including CHWs recruited from community-based organizations, into multiple aspects of the trial protocol. The investigators aim to recruit up to N=60 children with asthma randomized into intervention and control groups in a 1:1 ratio, conduct baseline assessments of indoor air quality and airway health, and collect repeated assessments of air quality and airway health during the three-month intervention period and after the trial concludes. Study findings will inform future approaches to integrate HEPA air cleaners into existing CHW asthma education programs in this and similar communities.

DETAILED DESCRIPTION:
Communities in proximity to airports face increased exposures to air pollution generated from both roadway and aircraft traffic. Exposure to particulate air pollution increases risk of an asthma exacerbation ("asthma attack") and, consequently, the possibility of an emergency room or urgent care visit. Puget Sound communities near flight paths have higher baseline rates of asthma and higher rates of asthma-related emergency room visits. For this study, the investigators will test whether an indoor air quality intervention involving HEPA air filtration units can address disparities in indoor air pollution and asthma health in neighborhoods around the Seattle Tacoma (SeaTac) International airport. Previous studies have reported benefits to deploying HEPA filters in indoor spaces, including improved air quality, as well as, reduced frequency of asthma symptoms and exacerbations, which can lead to urgent care visits and hospitalizations. However, it is unknown whether a similar intervention will be effective for children with asthma exposed to airport-related pollution, specifically.

Researchers with the University of Washington, Department of Environmental and Occupational Health Sciences, with experience in pediatric airway health, air pollution monitoring, methods for improving air quality, and epidemiology will conduct this work. They will assess the effectiveness of an indoor air quality intervention in reducing exposure to indoor pollutants and avoiding asthma symptom flare-ups for children with asthma living near SeaTac International airport.

To conduct this study, a sample of children referred to the Public Health - Seattle & King County (PHSKC) Community Health Worker (CHW) Asthma Program and their caregivers will be recruited. Enrolled children and caregivers will be followed for 3 months in the AAA research study before they begin the CHW Asthma Education Program. Each will be randomized to an intervention group, which involves indoor air filtration using a HEPA air filter unit, or a control group, which receives an air filtration unit that may not reduce PM2.5 and ultrafine particulates, types of pollution specific to air and road traffic. About 60 families will participate in total across the two-year study period (January 2024 through June 2025).

The primary research questions assessed in this study are A) Does adding a HEPA filter intervention to the existing asthma education program improve asthma outcomes? and B) Is there an indoor air quality benefit to using an indoor HEPA filter in the homes impacted by aircraft-related air pollution?

Currently, the Community Health Worker (CHW) Asthma Program provides a range of educational services, a green cleaning kit, a HEPA vacuum and mattress encapsulation materials. It does not provide a portable HEPA filter for the participant's home bedroom. The purpose of this project is to assess the added benefit of adding the HEPA unit to future asthma education program interventions.

Caregivers will complete weekly questionnaires to track the occurrence of asthma symptoms, a marker of asthma exacerbations, and health care utilization for asthma. Air quality inside and outside the homes will be monitored. When the study is completed, the investigators will determine whether families in the intervention group had better air quality and improved asthma symptoms during the follow-up period. These findings will be disseminated to the community with the help of the CHWs.

ELIGIBILITY:
Inclusion Criteria:

* Child is 6-12 years old with a health care provider-diagnosed asthma.
* Caregiver is comfortable in participating in all study activities in English (communicating with study staff by phone and completing online surveys).
* Caregiver is familiar with the child's daily asthma health.
* Residence within 10 miles of Seattle-Tacoma International Airport as determined by zip code
* Child resides in caregiver's home at least five nights a week on a regular basis and has no plans to move in the next three months.

Exclusion Criteria:

* Child has severe asthma at baseline. Severe asthma was defined in consultation with pediatric pulmonologists to be caregiver-reported asthma symptoms every day over the past 14 days and/or two or more inpatient hospitalizations for asthma in the past 12 months.
* Households were excluded if there were multiple individuals within the same household with asthma eligible for the King County CHW Asthma Program or had severe asthma.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Symptom days over 7 days | Repeated measure, assessed on a weekly basis throughout the 3 month observation period.
  Symptom days were assessed through brief weekly online surveys sent to caregivers. A symptom-day was defined as any day in the past week when the child had asthma symptoms or used quick-relief medication. Caregivers reported the number of days with symptoms (e.g., coughing, wheezing, shortness of breath, nighttime awakenings), any unscheduled medical visits, and whether the child had a respiratory infection. They also noted how many nights the child slept at home, any issues with the indoor air cleaner, and its usage frequency.
  Symptom scores ranged from 0 to 7, with high scores indicating more days experienced for that symptom.
  Study staff monitored the weekly caregiver survey to ensure that the child's symptoms were not worsening over the course of the study.
Change in Asthma Control Score | From the baseline visit until the end of study follow-up, 3 months later.
  The Child Asthma Control Test (C-ACT) is a short seven-question survey used to characterize child asthma control based on parent and child report of symptoms over the prior 30 days. The C-ACT has been validated for ages 4-11 years old and shown to have good psychometric properties. A C-ACT score is calculated based on responses, ranging from 0 to 27, with higher values reflecting better asthma control, and a score of 19 or lower considered to reflect inadequate, or "poor," control. This test is administered at the beginning and at the end of the research study. The change in child Asthma Control Test (C-ACT) score between baseline and post-intervention is used to assess the benefit of reducing indoor air pollution in the child's bedroom. Study team staff review responses on the baseline survey to address missing data or participant confusion during the study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Austin, Sc.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified information on indoor and outdoor air quality over the course of the study period will be shared through an open source publication. De-identified weekly symptom questionnaire will be shared, however identifiable participant information including age, gender/sex and home address will be redacted.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The study protocol, analysis plan is currently being prepared as an open-source publication to be shared with other researchers. The clinical study report and analytic code will be shared with researchers through open-source publication.
Access Criteria: A data management plan is available through dmptool.org allowing researchers to identify and request data elements that are not available through open source mechanisms.
URL: https://dmptool.org/plans/138914

REFERENCES:
- [Derived] Loftus CT, Lim P, Capps J, Shirai JH, Tchong-French M, Austin E. The Airport Air Quality and Asthma (AAA) indoor air intervention trial for children with asthma: Protocol for a community-based study in South King County, Washington State. Trials. 2025 Nov 27;26(1):596. doi: 10.1186/s13063-025-09286-8. PMID 41310837
- [Derived] Loftus C, Lim P, Capps J, Shirai J, Tchong-French M, Austin E. The Airport, Air Quality and Asthma (AAA) Indoor Air Intervention Trial for Children with Asthma: Protocol for a Community Based Study in South King County, Washington State. Res Sq [Preprint]. 2025 Sep 22:rs.3.rs-7181465. doi: 10.21203/rs.3.rs-7181465/v1. PMID 41041530
- See also: Project site detailing intervention design and planned phases. — https://deohs.washington.edu/aaa-study

DOCUMENTS (1):
  • Informed Consent Form (2024-02-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT07047430/ICF_000.pdf